CLINICAL TRIAL: NCT06370780
Title: Exploring, Predicting, and Intervening on Long-term Viral Suppression Electronically
Acronym: EPI-LoVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Florida State University (Other); University of California, Irvine (Other); University of North Carolina, Chapel Hill (Other); AIDS Healthcare Foundation (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Pamina Mae Gorbach, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-000477; 5UG3AI176592-02 (NIH)
Record Dates: First submitted 2024-04-10; First posted 2024-04-17 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Masking Description: N/A - all participants get the app
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Download the REMAIN App (Other): All participants download the app
  Interventions: Other: EPI LOVE

INTERVENTIONS:
Other: EPI LOVE — Observational cohort only

SUMMARY:
Despite the widespread availability of effective antiretroviral therapy (ART) in the United States, there remains significant numbers of people living with HIV (PLWH) who fail to achieve and or maintain viral suppression (VS). Disparities persist with the lowest levels of VS among Black individuals, people who use drugs, youth ages 18-24 and people residing in rural areas. Investigators will examine the syndemics underlying these outcomes including substance use, mental health, and barriers to HIV care including racial discrimination, stigma and rural isolation.

DETAILED DESCRIPTION:
This study will follow a digital cohort via the REMAIN App. The REMAIN App is adapted from the HealthMPowerment (HMP) platform and tailored to our focus population's unique needs. Digital cohorts, or eCohorts, utilize the flexibility and capacity of the internet to complement traditional approaches to epidemiological research, helping address some of the limitations and challenges associated with conventional cohort studies.

Aim 1 of this study is to recruit and retain a geographically and demographically diverse cohort of PLWH who are sub optimally engaged in care and with a history of, at high risk for, or not currently virally suppressed. Outcomes for this are levels of recruitment and retention to hit the study objectives to enroll 1,000 PLWH at risk for or experiencing VNS and follow them for up to 48 months. Aim 2 is to evaluate longitudinal patterns of care engagement within the cohort by modeling and advanced epidemiologic methods utilizing remote collection of biomarkers of HIV disease (e.g., viral load), online surveys, and brief, frequent app-based "check-ins". Outcomes include both those related to VS and engagement in care as well as engagement in the digital cohort.

ELIGIBILITY:
Inclusion Criteria:

* Have access to a personal smartphone device;
* Over 18 years of age;
* Speak English or Spanish;
* Living with HIV
* Are either 1) not currently virally suppressed, 2) not currently engaged in care, or 3) have one or more factors associated with viral non suppression including a history of missed appointments or viral non suppression;
* Active substance use or mental health disorder;
* Willing and able to provide written informed consent to take part in the study.

Exclusion Criteria:

* Unwilling or unable to provide reliable contact information;
* Unwilling to provide blood sample for HIV virology testing;
* Living with HIV and virally suppressed and not at risk of becoming unsuppressed in the near future.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of HIV Viral Suppression | past 3 months
  Suppression defined as having less than 200 copies of HIV per milliliter of blood.
Level of Adherence to HIV medication | past 6 months
  Adherence of at least 80% to ARV medication
Level of Adherence based on HIV appointments | one year
  Adherence defined as not missing more than 1 HIV care appointment in 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pamina Gorbach, DrPh, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States